CLINICAL TRIAL: NCT02229591
Title: Expiratory Flow Limitation and Postoperative Complications
Status: Completed | Type: Observational
Sponsor: Università degli Studi di Ferrara (Other)
Responsible Party: Principal Investigator, Savino Spadaro, Universitary Researcher, Università degli Studi di Ferrara
Other Study IDs: 17082014
Record Dates: First submitted 2014-08-28; First posted 2014-09-01 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Postoperative Respiratory Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- EFL patients: Patients with Expiratory Flow Limitation undergoing surgery
- Control group: Patients withouth Expiratory Flow Limitation undergoing surgery

SUMMARY:
Expiratory flow limitation (EFL) occurs when flow ceases to increase with increasing expiratory effort. In any circumstances EFL predisposes to pulmonary dynamic hyperinflation and its unfavorable effects such as increased elastic work of breathing, inspiratory muscles dysfunction, and progressive neuroventilatory dissociation, leading to reduced exercise tolerance, marked breathlessness during effort, and severe chronic dyspnea. Our hypothesis is that EFL should affect post operative outcomes like incidence of pulmonary complication and length of stay in hospital

ELIGIBILITY:
Inclusion Criteria:

* General anesthesia
* Duration of the surgery >2 hours

Exclusion Criteria:

* <18 years
* Consensus not given

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing abdominal, thyroid or vascular surgery in Sant'Anna Hospital
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2013-01; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Pulmonary complication | 28 days
  Postoperative pulmonary complication such infection, acute respiratory distress, post operative desaturation

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero Universitaria Sant'Anna, Ferrara, Italy